CLINICAL TRIAL: NCT06683976
Title: Safety and Efficacy of Improvised Chest Tube Drainage in the Absence of Conventional Systems: a Prospective Single-Center Study in Emergency and Conflict Zones in Sudan
Brief Title: Evaluating Improvised Chest Drainage Techniques in Conflict Zones
Status: Completed | Type: Observational
Sponsor: Sudan Medical Specialization Board (Other Government)
Responsible Party: Principal Investigator, Alsadig Suliman, Principal Investigator, Sudan Medical Specialization Board
Other Study IDs: WADMAD-ICDS-2024-01
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Pneumothorax; Hemothorax; Thoracic Trauma; Flail Chest; Hemopneumothorax; Traumatic
Keywords: Underwater Seal System Alternatives; Chest Trauma; Improvised Chest Drainage; Nasogastric Tube Chest Drain; Low-Resource Trauma Care; Conflict Zone Healthcare; Pneumothorax Management; Hemothorax Treatment; Alternative Chest Tube Methods; Emergency Thoracic Intervention
MeSH Terms: conditions — Pneumothorax; Hemothorax; Flail Chest; Hemopneumothorax; Thoracic Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard Treatment Group Label: Conventional Chest Drainage: This group includes patients with chest trauma who receive standard chest drainage using commercial chest tubes and underwater seal systems. This intervention follows established guidelines and protocols for chest drainage in trauma care. Patients in this group serve as the control group for comparing outcomes with those receiving improvised drainage systems.
- Improvised Treatment Group Label: Improvised NG Tube Drainage: This group includes patients with chest trauma who receive chest drainage using improvised methods, specifically nasogastric (NG) tubes as chest drains and intravenous (IV) drip sets adapted to function as underwater seals. This alternative intervention is used due to resource constraints and aims to evaluate the safety and effectiveness of improvised methods in a low-resource, conflict-affected setting

SUMMARY:
This study examines the use of improvised chest drainage systems in managing chest trauma at Wad Madani Teaching Hospital, a low-resource and conflict-affected setting. Due to a shortage of standard chest tubes and underwater seal systems, healthcare providers have adapted by using nasogastric (NG) tubes as chest drains and IV drip sets as makeshift underwater seals.

The study aims to evaluate the safety, effectiveness, and feasibility of these improvised methods compared to traditional chest drainage techniques. Primary outcomes will include lung re-expansion success, infection rates, and hospital stay length. By assessing patient outcomes, this study seeks to determine if these adapted techniques can provide a viable alternative for trauma care in resource-limited settings, potentially guiding practices in similar environments globally.

DETAILED DESCRIPTION:
This study explores the application of improvised chest drainage systems at Wad Manani Teaching Hospital for managing chest trauma in a low-resource, conflict-affected setting. Due to limited availability of standard medical supplies, an alternative approach has been adopted using nasogastric (NG) tubes as chest drains paired with intravenous (IV) drip sets, modified to act as underwater seals.

The primary aim is to assess the safety and effectiveness of these improvised systems in comparison to conventional chest tube drainage. By focusing on outcomes such as lung re-expansion success, infection rates, and recovery time, this study seeks to establish the clinical viability of improvised drainage systems in emergencies. Secondary evaluations include cost-effectiveness and the role of targeted staff training in improving procedural outcomes.

Study Approach:

This is a 6-months prospective observational study where patients with chest injuries are assigned to either a standard treatment group or an improvised treatment group. The improvised system involves inserting an NG tube as a chest drain connected to a modified IV drip set for underwater sealing. Standard sterile protocols are followed to reduce infection risk.

Data Collection & Analysis:

Data on each patient's clinical course and intervention will be recorded, focusing on primary outcomes like successful lung re-expansion and infection, and secondary outcomes, including procedural feasibility and cost. Comparative statistical analysis will assess outcome differences between groups.

Ethical Compliance:

Institutional review board (IRB) approval will be obtained, with all patient data anonymized and securely stored. Informed consent will be obtained from all participants or their guardians.

Impact Statement:

By assessing improvised methods in trauma care within a resource-limited context, this study could inform adaptable practices for similar environments worldwide, potentially influencing trauma care protocols and patient outcomes in challenging settings.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Patients presenting with chest trauma requiring chest drainage (e.g., pneumothorax, hemothorax)
* Willingness to provide informed consent to participate in the study -Stable enough to undergo chest X-ray or clinical assessment for lung re- expansion

Exclusion Criteria:

* Patients with pre-existing severe lung disease or significant comorbidities affecting chest drainage outcomes (e.g., advanced COPD, heart failure)
* Patients with prior chest surgery that may interfere with drainage outcomes
* Individuals with contraindications to chest tube insertion or NG tube placement
* Patients unwilling or unable to provide informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients (18 years and75 years) presenting with chest trauma at Wad Madani Teaching Hospital, a low-resource and conflict-affected setting. Patients are eligible if they require chest drainage for conditions such as pneumothorax or hemothorax and are stable enough to undergo the procedure. Due to limited resources, chest drainage methods include both standard and improvised techniques. The study population represents individuals receiving trauma care in a low-resource setting, providing insights into the effectiveness and safety of adapted drainage techniques in resource-constrained environments
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients With Successful Lung Re-expansion | Within 72 hours post-drainage
  The percentage of patients in each group (conventional vs. improvised chest drainage) who achieve full lung re-expansion as confirmed by chest X-ray.

SECONDARY OUTCOMES:
Rate of Drainage-Related Infections | Up to 30 days post-procedure
  Number of participants with infections directly associated with the chest drainage procedure, including pleural or wound infections, documented by clinical signs and laboratory findings.
Median Length of Hospital Stay | From admission to discharge (typically within 30 days)
  Median number of days from admission to discharge for each participant, allowing for the assessment of recovery duration associated with each drainage method.

OTHER OUTCOMES:
Patient Satisfaction Score at Discharge | At discharge (up to 30 days post-procedure)
  Patient satisfaction score assessed using a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied) at discharge, indicating the participant's perceived comfort and effectiveness of the chest drainage method used.

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Ali Musa, Consultant, Study Chair — University of Gezira, Faculty of medicine
Locations (1):
- Wad Madani teaching Hospital, Wad Madani, Al Jazirah, Sudan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly due to several considerations. First, the data includes sensitive personal health information, which must be protected to comply with privacy regulations and ethical standards. Additionally, the study is conducted in a low-resource setting, where data management and sharing capabilities may be limited. Ensuring the confidentiality and anonymity of participants is paramount, and sharing IPD could compromise these ethical obligations. Finally, the data will be used exclusively for the purpose of this study to inform clinical practice within the context of the local healthcare system, rather than for broader dissemination.